CLINICAL TRIAL: NCT06848192
Title: The Parkinson's Disease Case-Control Study: Gut Microbiome Study for Parkinson's Disease
Brief Title: The Parkinson's Disease Case-Control Study
Status: Recruiting | Type: Observational
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20250115ZJS001
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Blood (10 mL), stool sample (10 g), random midstream urine (12 mL)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Parkinson's Disease Case-Control Study is a study of healthy volunteers and patients with Parkinson's disease aged 50-75 years living in Hangzhou, China. This study aims to systematically investigate the differences in intestinal fungi between patients and healthy volunteers, find the key strains, and explore the molecular mechanism of Parkinson's disease with multi-omics data. Another aim of this study is to explore the association between intestinal fungi and brain structure and function from the perspective of the gut-brain axis by combining brain image data.

DETAILED DESCRIPTION:
Parkinson's disease is the second most common neurodegenerative disease of the central nervous system. Recent studies have shown that gut microorganisms, through their metabolites, can directly and indirectly affect brain function and neurodegenerative processes through the immune system, endocrine system, and nervous system, thus affecting the progress of Parkinson's disease. Gut fungi, as an important component of gut microorganisms, are rarely studied in Parkinson's disease. To systematically explore the differences in intestinal fungi between patients with Parkinson's disease and healthy volunteers, this project is expected to recruit 20 healthy volunteers and 20 Parkinson's disease patients respectively. The Parkinson's Disease Case-Control Study design incorporates collecting demographic information and clinical characteristics of Parkinson's disease patients and healthy volunteers, as well as biological samples (blood, urine, stool) and brain magnetic resonance imaging (MRI) of the subjects.

ELIGIBILITY:
Inclusion Criteria:

(For PD patients)

1. Men or women aged 50 to 75 years.
2. Clinical diagnosis of Parkinson's disease (based on MDS Parkinson's disease diagnostic criteria)
3. The patient must have at least two of the following symptoms: static tremor, bradykinesia, stiffness (which must include at least static tremor or bradykinesia); Or have asymmetrical resting tremors or asymmetrical bradykinesia.
4. Able to provide informed consent.

(For healthy volunteers)

1. Age (±2 years) and sex-matched healthy control individuals for each Parkinson's disease patient.
2. Able to provide informed consent.

Exclusion Criteria:

(For PD patients)

1. Atypical or secondary parkinsonism due to medications (e.g., metoclopramide, flunarizine, antipsychotics) or metabolic diseases (e.g., Wilson's disease), encephalitis, or degenerative diseases (e.g., progressive supranuclear palsy).
2. The presence of clinically diagnosed dementia as determined by the investigator.
3. Previous MRI scans showed clinically significant neurological disorders (as judged by the investigator).
4. Serious illness (e.g., heart failure or malignancy).
5. Smoking more than 15 cigarettes a day and a history of alcohol or drug addiction
6. Inflammatory gastrointestinal diseases.
7. Chronic diseases that may affect the gut microorganism (e.g., diabetes, cirrhosis, or cardiovascular disease).
8. Blood or autoimmune disease, or use of immunosuppressants in the past 3 months.
9. Antibiotics have been used within 3 months prior to sample collection.
10. Chronic constipation.

(For healthy volunteers)

1. Have a first-degree relative with Parkinson's disease (e.g. biological parent, sibling, or child).
2. Current or past clinically significant neurological disorders (as judged by the investigator).
3. Previous MRI scans showed clinically significant neurological disorders (as judged by the investigator).
4. Use of the following drugs in the 6 months prior to the screening visit: dopamine blockers (antipsychotics), metoclopramide, and riserpine.
5. Inflammatory gastrointestinal diseases.
6. Smoking more than 15 cigarettes a day and a history of alcohol or drug addiction
7. Chronic diseases that may affect the gut microorganism (e.g., diabetes, cirrhosis, or cardiovascular disease).
8. Blood or autoimmune disease, or use of immunosuppressants in the past 3 months.
9. Antibiotics have been used within 3 months prior to sample collection.
10. Chronic constipation.
11. Participating in other clinical trials

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the participants should be residents living in Hangzhou, China
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome profiling | At enrollment
  The microbiome profile is analyzed based on stool samples.

SECONDARY OUTCOMES:
Fecal and serum metabolomics profiling | At enrollment
  Metabolomics profiles are analyzed based on blood samples and stool samples.
Blood and urine proteomics profiling | At enrollment
  Proteomics profiles are analyzed based on blood samples and urine samples.
Brain imaging features | At enrollment
  MRI scans are used to extract brain imaging features.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided